CLINICAL TRIAL: NCT02683083
Title: Phase I Study to Evaluate the Safety, Biodistribution, Radiation Dosimetry and Tumor Imaging Potential of [131I]-SGMIB Anti-HER2 VHH1 in Healthy Volunteers and Breast Cancer Patients: CAM-VHH1 Study
Brief Title: Study to Evaluate the Safety, Biodistribution, Radiation Dosimetry and Tumor Imaging Potential of [131I]-SGMIB Anti-HER2 VHH1 in Healthy Volunteers and Breast Cancer Patients
Acronym: CAM-VHH1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Precirix (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CAM-VHH1; 2015-004840-21 (EudraCT Number)
Record Dates: First submitted 2016-02-09; First posted 2016-02-17 (Estimated); Results first posted 2019-07-18 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-07

CONDITIONS: Healthy Volunteers; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- [131I]-SGMIB Anti-HER2 VHH1 (Experimental)
  Interventions: Biological: [131I]-SGMIB Anti-HER2 VHH1

INTERVENTIONS:
Biological: [131I]-SGMIB Anti-HER2 VHH1

SUMMARY:
Primary purpose of the clinical study is to evaluate the safety, biodistribution and radiation dosimetry of [131I]-SGMIB Anti-HER2 VHH1 in healthy volunteers and patients with HER2+ breast cancer.

Secondary purpose of the clinical study is to evaluate the tumor uptake of [131I]-SGMIB Anti-HER2 VHH1 in patients with HER2+ breast cancer.

ELIGIBILITY:
Inclusion Criteria:

Subjects will only be included in the study if they meet all of the following criteria:

* Subjects who have given informed consent
* Subjects that agree not to drink alcoholic beverages or use any drugs during the study
* Subject with blood parameters within normal ranges
* Age: at least 18 years old

Patients will only be included in the study if they meet all of the following criteria:

* Patients who have given informed consent
* Patients that agree not to drink alcoholic beverages or use any drugs during the study
* Age: at least 18 years old
* Patients with local, locally advanced or metastatic HER2+ breast carcinoma as diagnosed on biopsied tissue by immunohistochemistry or fluorescence in situ hybridization (FISH).

Exclusion Criteria:

Patients will not be included in the study if one of the following criteria applies:

* Pregnant patients
* Breast feeding patients
* Patients with occupational exposure to ionizing irradiation
* Patients with previous thyroid disorders
* Patients that received radiolabeled compounds with a long half-life (>7h) for diagnostic or therapeutic purposes within the last 2 days.
* Patients with absolute contra-indications for thyroid blockage with potassium iodide.
* Patients with abnormal liver: ALT/AST > 2 times normal values; bilirubin > 1.5 time normal values.
* Patients with abnormal kidney function: < 50 ml/min/1,73 m2
* Patients with recent (< 1 week) gastrointestinal disorders (CTCAE v4.0 grade 3 or 4) with diarrhea as major symptom
* Patients with any serious active infection
* Patients who have any other life-threatening illness or organ system dysfunction, which in the opinion of the investigator would either compromise patient safety or interfere with the evaluation of the safety of the test radiopharmaceutical
* Patients who cannot communicate reliably with the investigator
* Patients who are unlikely to cooperate with the requirements of the study
* Patients at increased risk of death from a pre-existing concurrent illness
* Patients who participated already in this study
* Patients who participated in a previous trial with Anti-HER2 VHH1

Subjects will not be included in the study if one of the following criteria applies:

* Pregnant subjects
* Breast feeding subjects
* Subjects with occupational exposure to ionizing irradiation
* Subjects with clinical significant disease or on concomitant therapy (except contraception)
* Subjects with previous thyroid disorders
* Subjects that received radiolabeled compounds with a long half-life (>7h) for diagnostic or therapeutic purposes within the last 2 days.
* Subjects with absolute contra-indications for thyroid blockage with potassium iodide.
* Subjects with abnormal liver: ALT/AST > 2 times normal values; bilirubin > 1.5 time normal values.
* Subjects with abnormal kidney function: < 50 ml/min/1,73 m2
* Subjects with recent (< 1 week) gastrointestinal disorders (CTCAE v4.0 grade 3 or 4) with diarrhea as major symptom
* Subjects with any serious active infection
* Subjects who have any other life-threatening illness or organ system dysfunction, which in the opinion of the investigator would either compromise subject safety or interfere with the evaluation of the safety of the test radiopharmaceutical
* Subjects who cannot communicate reliably with the investigator
* Subjects who are unlikely to cooperate with the requirements of the study
* Subjects at increased risk of death from a pre-existing concurrent illness
* Subjects who participated already in this study
* Subjects who participated in a previous trial with Anti-HER2 VHH1

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-10; Primary Completion 2018-02-05 (Actual); Study Completion 2018-02-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Brussels, Choose A State, Belgium

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- [131I]-SGMIB Anti-HER2 VHH1: All subjects received one single intravenous injection of the investigational medical product ([131I]-SGMIB Anti-HER2 VHH1).
Period: Overall Study
Arm/Group | [131I]-SGMIB Anti-HER2 VHH1
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | [131I]-SGMIB Anti-HER2 VHH1
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.78 (18.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v4.0
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | [131I]-SGMIB Anti-HER2 VHH1
Number analyzed (Participants) | 9
Participants | 0

2. Secondary Outcome: The Tumor Targeting Potential Will be Visually Scored on the Planar Total Body Scan
Description: Cancer lesions above 3 cm will be visually interpreted by an experienced nuclear medicine physician. Lesions will be scored positive if CAM-H2 uptake in the lesion is higher than surrounding background.
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | [131I]-SGMIB Anti-HER2 VHH1
Number analyzed (Participants) | 3
Participants | 2

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | [131I]-SGMIB Anti-HER2 VHH1
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 4/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | [131I]-SGMIB Anti-HER2 VHH1 (N=9)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Adhesive plaster sensitivity (Skin and subcutaneous tissue disorders) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-04): https://cdn.clinicaltrials.gov/large-docs/83/NCT02683083/Prot_SAP_000.pdf